CLINICAL TRIAL: NCT06891872
Title: Immunogenicity and Safety of Live Attenuated Varicella Vaccine Co-administered with MMR Vaccine or DTaP Vaccine in Healthy Children Aged 18~24 Months: an Open-label, Randomized, Phase Ⅳ Study Clinical Trial
Brief Title: Study of Live Attenuated Varicella Vaccine Co-administered with MMR Vaccine or DTaP Vaccine
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac (Dalian) Vaccine Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO-VZV-4008
Record Dates: First submitted 2025-03-02; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Varicella (chickenpox); MMR Vaccine; DTaP Vaccine
Keywords: Co-administered; VZV
MeSH Terms: conditions — Chickenpox | interventions — Chickenpox Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Varicella vaccine and DTaP co-administration group ) (Experimental): Participants will receive a single dose of varicella vaccine and DTaP vaccine on Day 0 and a single dose of MMR on Day 30.
  Interventions: Biological: Vaicella Vaccine+DTaP on Day 0, MMR on Day 30
- Group B (Varicella vaccine and MMR co-administration group ) (Experimental): Participants will receive a single dose of varicella vaccine and MMR on Day 0 and DTaP vaccine on Day 30.
  Interventions: Biological: Varicella vaccine+MMR on Day 0，DTaP on Day 30
- Group C (Varicella vaccine group ) (Active Comparator): Participants will receive a single dose of varicella vaccine on Day 0.
  Interventions: Biological: Varicella Vaccine

INTERVENTIONS:
Biological: Vaicella Vaccine+DTaP on Day 0, MMR on Day 30 — Varicella vaccine: lyophilized powder, subcutaneous injection
  DTaP: intramuscular injection
  MMR: lyophilized powder, subcutaneous injection
  Arms: Group A (Varicella vaccine and DTaP co-administration group )
Biological: Varicella vaccine+MMR on Day 0，DTaP on Day 30 — Varicella vaccine: lyophilized powder, subcutaneous injection
  MMR: lyophilized powder, subcutaneous injection
  DTaP: intramuscular injection
  Arms: Group B (Varicella vaccine and MMR co-administration group )
Biological: Varicella Vaccine — lyophilized powder, subcutaneous injection
  Arms: Group C (Varicella vaccine group )

SUMMARY:
This is a phase Ⅳ clinical trial of live attenuated varicella vaccine manufactured by Sinovac (Dalian) Vaccine Technology Co., Ltd.The primary objective of this study is to evaluate the immunogenicity of live attenuated varicella vaccine co-administered with MMR vaccine or DTaP vaccine. The secondary objective is to evaluate the safety of the vaccines when administered simultaneously.

DETAILED DESCRIPTION:
A total of 720 children aged 18~24 months who have not received varicella vaccine, the second dose of MMR and the fourth dose of DTaP (or vaccines containing related ingredients) will be recruited and randomly assigned to one of three study groups (1:1:1 ratio): Group A, Group B and Group C. Participants in Group A will receive varicella vaccine and DTaP simultaneously on Day 0 and receive MMR on Day 30. Participants in Group B will varicella vaccine and MMR simultaneously on Day 0 and receive DTaP on Day 30. Participants in Group C will receive varicella vaccine only.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged 18-24 months;
* have completed 3 doses of DTaP for primary immunization in their first year of life without the fourth dose of Dtap-containing vaccine;
* have completed the first dose of MMR in their first year of life without a second dose of MMR;
* Guardians of participants who are able to understand and voluntarily sign informed consent;
* Provision of legal proof of identity.

Exclusion Criteria:

* Having a history of previous varicella vaccination;
* Having a history of chickenpox, pertussis, diphtheria, tetanus, measles, mumps, and rubella;
* Having a history of uncontrolled chronic or serious diseases, including but not limited to cardiovascular diseases, hematological diseases, liver and kidney diseases, digestive diseases, respiratory diseases, malignant tumors, major functional organ transplantation, etc.;
* Presence of autoimmune diseases, immunodeficiency diseases (including but not limited to systemic lupus erythematosus, ankylosing spondylitis, autoimmune thyroid disease, asplenia, functional asplenia, HIV infection);
* Presence of abnormal coagulation function (e.g. coagulation factor deficiency, platelet abnormality);
* Having/Previous having a severe neurological disorder (epilepsy, seizures, or convulsions) or psychosis, or have a family history of psychosis;
* Acute onset of various acute or chronic illnesses within the last 7 days, or known or suspected active infection;
* Receipt of > 14 days of immunosuppressive or other immunomodulatory therapy (prednisone ≥2 mg/kg/ day or its equivalent, except topical or inhaled corticosteroids), cytotoxic therapy within the past 6 months, or planned to receive such therapy during the trial;
* Having received immune globulin or other blood products within the past 3 months or plan to receive such treatment during the trial;
* Receipt of another study drug or vaccine within the past 30 days or plans to receive such drug or vaccine during the trial;
* Administration of live attenuated vaccine within the past 28 days or subunit, inactivated, or other process vaccine within the past 7 days;
* Known allergies to the vaccine or vaccine components, such as urticaria after vaccination, dyspnea, angioedema;
* Having fever on the day of scheduled vaccination (axillary temperature > 37.0 ° C);
* Failure of medical examination on the planned vaccination day;
* Participants have any other factors that, in the judgment of the investigator, make them ineligible to participate in a clinical trial.

Ages: 18 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 720 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Varicella zoster virus (VZV) antibody seroconversion rate | Day 30 after the administration of varicella vaccine
  Seroconversion rate of VZV antibody on Day 30 after the administration of varicella vaccine.

SECONDARY OUTCOMES:
Seropositive rate of VZV antibody | Day 30 after the administration of varicella vaccine
  Seropositive rate of VZV antibody on Day 30 after the administration of varicella vaccine.
Geometric mean titer (GMT) of VZV antibody | Day 30 after the administration of varicella vaccine
  GMT of VZV antibody on Day 30 after the administration of varicella vaccine.
Geometric mean fold increase (GMI) of VZV antibody | Day 30 after the administration of varicella vaccine
  GMI of VZV antibody on Day 30 after the administration of varicella vaccine.
Seroconversion rate of measles antibody, mumps antibody and rubella antibody | Day 30 after the administration of MMR
  Seroconversion rate of measles antibody, mumps antibody and rubella antibody on Day 30 after the administration of MMR
Seropositive rate of measles antibody, mumps antibody and rubella antibody | Day 30 after the administration of MMR
  Seropositive rate of measles antibody, mumps antibody and rubella antibody on Day 30 after the administration of MMR
Geometric mean concentration (GMC) of measles antibody, mumps antibody and rubella antibody | Day 30 after the administration of MMR
  GMC of measles antibody, mumps antibody and rubella antibody on Day 30 after the administration of MMR
GMI of measles antibody, mumps antibody and rubella antibody | Day 30 after the administration of MMR
  GMI of measles antibody, mumps antibody and rubella antibody on Day 30 after the administration of MMR
Seroconversion rate of pertussis antibody, diphtheria antibody and tetanus antibody | Day 30 after the administration of DTaP
  Seroconversion rate of pertussis antibody, diphtheria antibody and tetanus antibody on Day 30 after the administration of DTaP
Seropositive rate of pertussis antibody, diphtheria antibody and tetanus antibody | Day 30 after the administration of DTaP
  Seropositive rate of pertussis antibody, diphtheria antibody and tetanus antibody on Day 30 after the administration of DTaP
GMC of pertussis antibody, diphtheria antibody and tetanus antibody | Day 30 after the administration of DTaP
  GMC of pertussis antibody, diphtheria antibody and tetanus antibody on Day 30 after the administration of DTaP
GMI of pertussis antibody, diphtheria antibody and tetanus antibody | Day 30 after the administration of DTaP
  GMI of pertussis antibody, diphtheria antibody and tetanus antibody on Day 30 after the administration of DTaP
The incidence of adverse reactions within 0~14 days | 0~14 days after each dose vaccination
  The incidence of adverse reactions within 0~14 days after each dose vaccination.
The incidence of adverse reactions within 0~30 days | 0~30 days after each dose vaccination
  The incidence of adverse reactions within 0~30 days after each dose vaccination.
The incidence of serious adverse events (SAEs) within 0~30 days | 0~30 days after each dose vaccination
  The incidence of SAEs within 0~30 days after each dose vaccination.

CONTACTS AND LOCATIONS:
Locations (1):
- Chongqing Center for Disease Control and Prevention, Chongqing, China

IPD SHARING:
Plan to Share IPD: No